CLINICAL TRIAL: NCT05741840
Title: Telehealth Parent-only Treatment for Youth With Autism Spectrum Disorder and Overweight/Obesity
Brief Title: Family, Responsibility, Education, Support, and Health for Families With a Child With Autism
Acronym: FRESH-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Kerri Boutelle, Professor of Pediatrics, Psychiatry, and Herbert Wertheim School of Public Health and Human Longevity Science, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 802230; R01HD106991 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder; Obesity, Childhood; Autism
Keywords: obesity; treatment; intervention; Autism; behavioral treatment; parent based treatment; children
MeSH Terms: conditions — Autism Spectrum Disorder; Pediatric Obesity; Autistic Disorder; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBT-A (Experimental): PBT-A includes the elements of family based behavioral treatment for children with obesity, delivered exclusively to a parent via telehealth.
  Interventions: Behavioral: PBT-A
- Health Education (Active Comparator): This program provides information about nutrition, physical activity, sedentary behavior, sleep, emotions, and stress delivered exclusively to a parent via telehealth.
  Interventions: Behavioral: Health Education (HE)

INTERVENTIONS:
Behavioral: PBT-A — PBT-A provides all the elements of family based treatment for children with obesity, including nutrition and physical activity education, behavior therapy skills, and parenting skills.
  Other Names: parent based treatment; family based behavioral treatment
  Arms: PBT-A
Behavioral: Health Education (HE) — The HE arm will provide information about nutrition, physical activity, sedentary behavior, sleep, emotions, and stress.
  Arms: Health Education

SUMMARY:
The objective of this proposed study is to collect initial efficacy data on a telehealth parent-based behavioral program for children with autism and overweight or obesity (PBT-A), compared with health education (HE).

DETAILED DESCRIPTION:
The study will compare the efficacy of PBT-A and health education program delivered via telehealth to parents on child weight management. Investigators will provide 6 months of a group program (PBT-A or HE) and will follow participants for 12-months post-treatment (total time = 18 months). Investigators will recruit parents of children diagnosed with autism and overweight or obesity. Assessments will occur at 5 timepoints: baseline, mid-treatment, post-treatment, 6-month and 12-month follow-up. Assessments will include anthropometry for both parent and child. Parent will also provide information regarding autism diagnosis and characteristics, eating behaviors, and parenting relationship measures. This program of research has the potential to advance the standard of practice for children with autism and overweight or obesity by developing tailored interventions which can be easily disseminated.

ELIGIBILITY:
Inclusion Criteria:

1. A child with OW/OB (>=85% BMI for age) aged 6-12 years
2. Documented (1) community diagnosis or provisional diagnosis of ASD or (2) educational diagnosis of ASD
3. The child meets cut-off criteria for autism on the Autism Diagnostic Interview-Revised (ADI-R), as well as overall DSM 5 criteria based on the clinical judgement of an experienced clinician
4. The parent who is responsible for food preparation is willing to participate
5. The family is willing to commit to attending all treatment and assessment sessions
6. Child on a stable regimen of prescription medications which affect appetite or weight (minimum of 3 months)
7. Child does not have any medical conditions that limit ability to participate in physical activity for the duration of the study. Parent can participate in physical activity or at least facilitate support of child's completion of recommended physical activity.
8. Child and/or parent are not participating in another organized weight control program
9. Family owns a device that can facilitate zoom meetings

Exclusion Criteria:

1. Child diagnoses of a serious chronic physical disease (e.g., cystic fibrosis, type 1 diabetes) for which physician supervision of diet and/or exercise is needed
2. Child or first degree relative with diagnosis of anorexia or bulimia nervosa based on parent report
3. Acute parent psychiatric disorder (e.g., acute suicidality; recent hospitalization; psychosis, moderate or severe alcohol or substance use disorder) that could interfere with treatment.
4. Parent is not currently pregnant, lactating or planning to get pregnant during the study duration
5. Parent has had bariatric surgery less than 6 months ago and/or is not yet eating solid food or is planning to have bariatric surgery over the study duration
6. Child is taking medication for the purpose of weight loss

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Child BMIz age and sex adjusted BMI (kg/m^2) | Change from baseline to month 3, 6, 12, and 18
  age and sex adjusted body mass index (BMI) z-score based on the CDC norms
Child %BMIp95 | Change from baseline to month 3, 6, 12, and 18
  Age and Sex specific percentage of the 95th percentile BMI for age and sex that is more sensitive to change in children with higher weights

SECONDARY OUTCOMES:
Parent Dietary Intake | Change from baseline to month 6, 12, and 18
  Block Fat/Sugar/Fruit/Vegetable Screener for adults
Child Dietary Intake | Change from baseline to month 6, 12, and 18
  BLOCK kids food screener completed by parent
Parent Physical Activity | Change from baseline to month 6, 12, and 18
  The International Physical Activity Questionnaire (IPAQ)
Child Physical Activity | Change from baseline to month 6, 12, and 18
  The Children's Physical Activity Questionnaire (C-PAQ) parent proxy
Child Mealtime Behaviors | Change from baseline to month 6, 12, and 18
  The Brief Autism Mealtime Behavior Inventory (BAMBI) with scores ranging from 18 to 90 with higher scores indicating greater mealtime problem behaviors
Parent self-efficacy | Change from baseline to month 6, 12, and 18
  The Parenting Sense of Competence Scale (PSOC) - Scores range from 17-102 with higher scores representing higher parenting sense of competence.
Parent body mass index (BMI) | Change from baseline to mid-treatment, months: 3, 6, 12, and 18
  kg/m^2
Parenting as measured by the Alabama Parenting Questionnaire (APQ) | Change from baseline to month 6, 12, and 18
  Parents will self-report parenting behaviors via the APQ across 5 domains: 1) positive involvement with children, 2) supervision and monitoring, 3) use of positive discipline techniques, 4) consistency in the use of such discipline, and 5) use of corporal punishment. Higher scores indicate greater frequency of engagement with that particular parenting domain. Scores range from 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States